CLINICAL TRIAL: NCT03720327
Title: Fitness Intensive Therapy (Get FIT) to Promote Healthy Living in Older Adults
Brief Title: The Effects of a Mobile Health Intervention and Health Coach Text Messaging on Cardiovascular Risk of Older Adults
Acronym: GET FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Lorraine Evangelista, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: R21AG053162; HS#2016-2713; R21AG053162 (NIH)
Record Dates: First submitted 2018-10-09; First posted 2018-10-25 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two groups for the study duration (3 months):
  1. control group (Get FIT);
  2. intervention group (Get FIT+).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Get FIT (Active Comparator): The Get FIT intervention
  Interventions: Behavioral: Get FIT
- Get FIT+ (Experimental): The Get FIT+ intervention, which includes push-only personalized text messages from a health coach.
  Interventions: Behavioral: Get FIT+

INTERVENTIONS:
Behavioral: Get FIT — The Get FIT arm includes use of a free commercially available smartphone application to track daily food intake for 3 months; use of a Fitbit activity tracker for 3 months; and one 45 minute behavioral counseling session to set personal goals and provide education by a health coach.
  Arms: Get FIT
Behavioral: Get FIT+ — The Get FIT+ arm includes use of a free commercially available smartphone application to track daily food intake for 3 months; use of a Fitbit activity tracker for 3 months; one 45 minute behavioral counseling session to set personal goals and provide education by a health coach; and personalized text messaging for 3 months by a health coach. The health coach will have access to these participants' daily food and activity data through the smartphone application, and will monitor progress and send push-only text messages to participants in this group based on the participant's goals and progress in the areas of physical activity, nutrition, and weight loss.
  Arms: Get FIT+

SUMMARY:
This study, "Fitness Intensive Therapy (Get FIT) to Promote Healthy Living in Older Adults", will test a mobile-health based intervention which includes use of a Fitbit activity tracker for 3 months, a smartphone application that tracks daily food intake, and one 45 minute counseling session to create personal goals and provide patient education by a health coach; versus Get FIT+ (the same items) plus personalized text messages focusing on participant's activity and nutrition progress as monitored in the app, from the health coach for 3 months. The investigators will measure the impact on participant's diet, physical activity, clinical outcomes, psychosocial well-being, and engagement.

DETAILED DESCRIPTION:
This study, "Fitness Intensive Therapy (Get FIT) to Promote Healthy Living in Older Adults", will test 2 behavioral interventions in community-dwelling older adults (age ≥ 60 years) at intermediate and high risk of cardiovascular disease.

1. Get FIT: use of a Fitbit activity tracker, smartphone application to track daily food intake, one 45 minute counseling session to create personal goals and provide patient education by a health coach; vs.
2. Get FIT+: use of a Fitbit activity tracker, smartphone application to track daily food intake, one 45 minute counseling session to create personal goals and provide patient education by a health coach, and personalized push-only text messages from the health coach based on participant's progress as monitored electronically in the application.

Each intervention lasts 3 months, with outcomes measured at baseline, 3 months, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 or greater
* at intermediate (10-20%) or high risk (>20%) of developing cardiovascular disease (as measured by Framingham Risk Assessment Tool)
* poor eating behaviors (as measured by Block Fruit/Vegetable/Fiber Screener)
* reduced physical activity (as measured by Block Adult Physical Activity Screener)

Exclusion Criteria:

* cognitive impairment (as measured by Mini-Cog) that impairs ability to understand consent process, surveys, or use of mobile health devices
* chronic drug use
* end stage renal, liver, or pulmonary disease
* current active cancer (i.e., undergoing active treatment for cancer)
* gastrointestinal disease which requires a special diet (e.g. Crohn's, celiac, etc).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2022-03-12 (Actual); Study Completion 2022-03-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline adherence to recommended self-care behaviors at 3 months and 6 months | baseline, 3 months, 6 months
  The Medical Outcomes Study Specific Adherence Scale measures patient adherence to 8 recommended health behaviors (3 items on specific diet/nutrition, 1 item on smoking cessation, 1 item on alcoholic beverages, 1 item on taking prescribed medications, 1 item on regular exercise, 1 item on weight/fluid, 1 item on symptom management). Participants circle the answer that best corresponds to their behavior in the last 4 weeks ("None of the time; 1-A little of the time; 2-Some of the time; 3-A good bit of the time; 4-Most of the time; 5-All of the time"). Scoring is the average of the items for a total specific adherence score.
Change from Baseline diet patterns at 3 months and 6 months | baseline, 3 months, 6 months
  3-Day Food Record (ASA24); data from self-recorded diet as entered in smartphone application (My Fitness Pal©)
Change from baseline physical activity levels at 3 months and 6 months | baseline, 3 months, 6 months
  data from Fitbit activity tracker as recorded in smartphone application (My Fitness Pal©)

SECONDARY OUTCOMES:
change from baseline in HgA1c | baseline, 3 months, 6 months
  HgA1c as obtained by venous puncture and blood analysis
Change from baseline in Anxiety and Depression symptoms | baseline, 3 months, 6 months
  Anxiety and depression symptoms as measured by the Hospital Anxiety and Depression Scale (HADS). Subscale scores of Anxiety (range 0-21; lower scores representing "normal" scores) and Depression (range 0-21; lower scores representing "normal" scores).
Change from baseline in patient activation | baseline, 3 months, 6 months
  Patient activation as measured by the Patient Activation Measure
Change from Baseline height in centimeters | baseline, 3 months, 6 months
  height in centimeters as measured by stadiometer
Change from baseline weight in kilograms | baseline, 3 months, 6 months
  weight in kilograms as measured by professional beam scale
Change from baseline body composition-area | baseline, 6 months
  body composition-area (cm2) as measured by dual-energy x-ray absorptiometry (DEXA)
Change from baseline body composition-Bone Mineral Content (BMC) | baseline, 6 months
  body composition - BMC (g) as measured by dual-energy x-ray absorptiometry (DEXA)
Change from baseline body composition-Bone Mineral Density (BMD) | baseline, 6 months
  body composition - BMD (g/cm2) as measured by dual-energy x-ray absorptiometry (DEXA)
Change from baseline body composition-Fat mass | baseline, 6 months
  body composition - fat mass (g) as measured by dual-energy x-ray absorptiometry (DEXA)
Change from baseline body composition-Lean mass | baseline, 6 months
  body composition - lean mass (g) as measured by dual-energy x-ray absorptiometry (DEXA)
Change from baseline body composition-Total Mass | baseline, 6 months
  body composition - total mass (g) as measured by dual-energy x-ray absorptiometry (DEXA)
Change from baseline body composition-% fat | baseline, 6 months
  body composition - % fat as measured by dual-energy x-ray absorptiometry (DEXA)
Change from baseline in blood pressure | baseline, 3 months, 6 months
  blood pressure as measured by calibrated aneroid sphygmomanometer
Change from baseline in High-Density Lipoproteins (HDL) | baseline, 3 months, 6 months
  HDL as obtained by venous puncture and blood analysis
Change from baseline in Low-Density Lipoproteins (LDL) | baseline, 3 months, 6 months
  LDL as obtained by venous puncture and blood analysis
Change from baseline in Triglycerides | baseline, 3 months, 6 months
  Triglycerides as obtained by venous puncture and blood analysis
Change from baseline in total cholesterol score | baseline, 3 months, 6 months
  total cholesterol score as obtained by venous puncture and blood analysis (HDL+LDL+0.2*triglycerides=total)
change from baseline in quality of life | baseline, 3 months, 6 months
  quality of life as measured by the Quality of Life Short Form version 20
change from baseline in patterns of use of clinic attendance | baseline, 3 months, 6 months
  patient patterns of use as measured by clinic attendance
change from baseline in patterns of use of mHealth | baseline, 3 months, 6 months
  patient patterns of use as measured by use of mHealth
change from baseline in patterns of use of Retention | baseline, 3 months, 6 months
  patient patterns of use and engagement as measured by Retention (drop out rate and time of drop out)
cost effectiveness | 6 months
  Cost effectiveness of the intervention as calculated by the sum of costs of training, staff salary, frequency/duration of counseling sessions, follow up visits, real time feedback

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine Evangelista, PhD, Principal Investigator — University of California, Irvine
Locations (5):
- United States (5):
  - University of California, Irvine Federally Qualified Health Clinic, Anaheim, California
  - The Regents of the University of California, Irvine - Institute for Clinical & Translational Science (ICTS), Irvine, California
  - University of California, Irvine Medical Clinic (Gottschalk), Irvine, California
  - The University of California, Irvine Medical Center, Orange, California
  - University of California, Irvine Federally Qualified Health Clinic, Santa Ana, California

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Demiris G, Thompson H, Boquet J, Le T, Chaudhuri S, Chung J. Older adults' acceptance of a community-based telehealth wellness system. Inform Health Soc Care. 2013 Jan;38(1):27-36. doi: 10.3109/17538157.2011.647938. Epub 2012 May 9. PMID 22571733
- [Background] Schneider KM, O'Donnell BE, Dean D. Prevalence of multiple chronic conditions in the United States' Medicare population. Health Qual Life Outcomes. 2009 Sep 8;7:82. doi: 10.1186/1477-7525-7-82. PMID 19737412
- [Background] WRITING GROUP MEMBERS; Lloyd-Jones D, Adams RJ, Brown TM, Carnethon M, Dai S, De Simone G, Ferguson TB, Ford E, Furie K, Gillespie C, Go A, Greenlund K, Haase N, Hailpern S, Ho PM, Howard V, Kissela B, Kittner S, Lackland D, Lisabeth L, Marelli A, McDermott MM, Meigs J, Mozaffarian D, Mussolino M, Nichol G, Roger VL, Rosamond W, Sacco R, Sorlie P, Roger VL, Thom T, Wasserthiel-Smoller S, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2010 update: a report from the American Heart Association. Circulation. 2010 Feb 23;121(7):e46-e215. doi: 10.1161/CIRCULATIONAHA.109.192667. Epub 2009 Dec 17. No abstract available. PMID 20019324
- [Background] Lin JS, O'Connor E, Whitlock EP, Beil TL. Behavioral counseling to promote physical activity and a healthful diet to prevent cardiovascular disease in adults: a systematic review for the U.S. Preventive Services Task Force. Ann Intern Med. 2010 Dec 7;153(11):736-50. doi: 10.7326/0003-4819-153-11-201012070-00007. PMID 21135297
- [Background] Parekh AK, Goodman RA, Gordon C, Koh HK; HHS Interagency Workgroup on Multiple Chronic Conditions. Managing multiple chronic conditions: a strategic framework for improving health outcomes and quality of life. Public Health Rep. 2011 Jul-Aug;126(4):460-71. doi: 10.1177/003335491112600403. PMID 21800741
- [Background] Bodenheimer T, Wagner EH, Grumbach K. Improving primary care for patients with chronic illness: the chronic care model, Part 2. JAMA. 2002 Oct 16;288(15):1909-14. doi: 10.1001/jama.288.15.1909. PMID 12377092
- [Background] Kouris I, Mougiakakou S, Scarnato L, Iliopoulou D, Diem P, Vazeou A, Koutsouris D. Mobile phone technologies and advanced data analysis towards the enhancement of diabetes self-management. Int J Electron Healthc. 2010;5(4):386-402. doi: 10.1504/IJEH.2010.036209. PMID 21041177
- [Background] Chomutare T, Fernandez-Luque L, Arsand E, Hartvigsen G. Features of mobile diabetes applications: review of the literature and analysis of current applications compared against evidence-based guidelines. J Med Internet Res. 2011 Sep 22;13(3):e65. doi: 10.2196/jmir.1874. PMID 21979293
- [Background] Courtney KL, Demiris G, Rantz M, Skubic M. Needing smart home technologies: the perspectives of older adults in continuing care retirement communities. Inform Prim Care. 2008;16(3):195-201. doi: 10.14236/jhi.v16i3.694. PMID 19094406
- [Background] Hayes DK, Denny CH, Keenan NL, Croft JB, Sundaram AA, Greenlund KJ. Racial/Ethnic and socioeconomic differences in multiple risk factors for heart disease and stroke in women: behavioral risk factor surveillance system, 2003. J Womens Health (Larchmt). 2006 Nov;15(9):1000-8. doi: 10.1089/jwh.2006.15.1000. PMID 17125418
- [Background] Ford ES, Ajani UA, Croft JB, Critchley JA, Labarthe DR, Kottke TE, Giles WH, Capewell S. Explaining the decrease in U.S. deaths from coronary disease, 1980-2000. N Engl J Med. 2007 Jun 7;356(23):2388-98. doi: 10.1056/NEJMsa053935. PMID 17554120
- [Background] Maruthur NM, Wang NY, Appel LJ. Lifestyle interventions reduce coronary heart disease risk: results from the PREMIER Trial. Circulation. 2009 Apr 21;119(15):2026-31. doi: 10.1161/CIRCULATIONAHA.108.809491. Epub 2009 Apr 6. PMID 19349322
- [Background] Appel LJ, Brands MW, Daniels SR, Karanja N, Elmer PJ, Sacks FM; American Heart Association. Dietary approaches to prevent and treat hypertension: a scientific statement from the American Heart Association. Hypertension. 2006 Feb;47(2):296-308. doi: 10.1161/01.HYP.0000202568.01167.B6. PMID 16434724
- [Background] Elmer PJ, Obarzanek E, Vollmer WM, Simons-Morton D, Stevens VJ, Young DR, Lin PH, Champagne C, Harsha DW, Svetkey LP, Ard J, Brantley PJ, Proschan MA, Erlinger TP, Appel LJ; PREMIER Collaborative Research Group. Effects of comprehensive lifestyle modification on diet, weight, physical fitness, and blood pressure control: 18-month results of a randomized trial. Ann Intern Med. 2006 Apr 4;144(7):485-95. doi: 10.7326/0003-4819-144-7-200604040-00007. PMID 16585662
- [Background] Yusuf S, Hawken S, Ounpuu S, Dans T, Avezum A, Lanas F, McQueen M, Budaj A, Pais P, Varigos J, Lisheng L; INTERHEART Study Investigators. Effect of potentially modifiable risk factors associated with myocardial infarction in 52 countries (the INTERHEART study): case-control study. Lancet. 2004 Sep 11-17;364(9438):937-52. doi: 10.1016/S0140-6736(04)17018-9. PMID 15364185
- [Background] Kottke TE, Faith DA, Jordan CO, Pronk NP, Thomas RJ, Capewell S. The comparative effectiveness of heart disease prevention and treatment strategies. Am J Prev Med. 2009 Jan;36(1):82-88. doi: 10.1016/j.amepre.2008.09.010. PMID 19095166
- [Background] Svetkey LP, Erlinger TP, Vollmer WM, Feldstein A, Cooper LS, Appel LJ, Ard JD, Elmer PJ, Harsha D, Stevens VJ. Effect of lifestyle modifications on blood pressure by race, sex, hypertension status, and age. J Hum Hypertens. 2005 Jan;19(1):21-31. doi: 10.1038/sj.jhh.1001770. PMID 15385946
- [Background] Hall AK, Stellefson M, Bernhardt JM. Healthy Aging 2.0: the potential of new media and technology. Prev Chronic Dis. 2012;9:E67. Epub 2012 Mar 8. No abstract available. PMID 22405474
- [Background] Webb TL, Joseph J, Yardley L, Michie S. Using the internet to promote health behavior change: a systematic review and meta-analysis of the impact of theoretical basis, use of behavior change techniques, and mode of delivery on efficacy. J Med Internet Res. 2010 Feb 17;12(1):e4. doi: 10.2196/jmir.1376. PMID 20164043
- [Background] Osborn CY, Egede LE. Validation of an Information-Motivation-Behavioral Skills model of diabetes self-care (IMB-DSC). Patient Educ Couns. 2010 Apr;79(1):49-54. doi: 10.1016/j.pec.2009.07.016. Epub 2009 Aug 21. PMID 19699601
- [Background] Jaja C, Pares-Avila J, Wolpin S, Berry D. Usability evaluation of the interactive Personal Patient Profile-Prostate decision support system with African American men. J Natl Med Assoc. 2010 Apr;102(4):290-7. doi: 10.1016/s0027-9684(15)30601-5. PMID 20437736
- [Background] Moser DK, Dickson V, Jaarsma T, Lee C, Stromberg A, Riegel B. Role of self-care in the patient with heart failure. Curr Cardiol Rep. 2012 Jun;14(3):265-75. doi: 10.1007/s11886-012-0267-9. PMID 22437374
- [Background] Riegel B, Lee CS, Dickson VV; Medscape. Self care in patients with chronic heart failure. Nat Rev Cardiol. 2011 Jul 19;8(11):644-54. doi: 10.1038/nrcardio.2011.95. PMID 21769111
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564
- [Background] Dracup K, Evangelista LS, Hamilton MA, Erickson V, Hage A, Moriguchi J, Canary C, MacLellan WR, Fonarow GC. Effects of a home-based exercise program on clinical outcomes in heart failure. Am Heart J. 2007 Nov;154(5):877-83. doi: 10.1016/j.ahj.2007.07.019. Epub 2007 Sep 12. PMID 17967593
- [Background] Arean PA, Alvidrez J, Nery R, Estes C, Linkins K. Recruitment and retention of older minorities in mental health services research. Gerontologist. 2003 Feb;43(1):36-44. doi: 10.1093/geront/43.1.36. PMID 12604744
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Borson S, Scanlan J, Brush M, Vitaliano P, Dokmak A. The mini-cog: a cognitive 'vital signs' measure for dementia screening in multi-lingual elderly. Int J Geriatr Psychiatry. 2000 Nov;15(11):1021-7. doi: 10.1002/1099-1166(200011)15:113.0.co;2-6. PMID 11113982
- [Background] Parker C, Philp I. Screening for cognitive impairment among older people in black and minority ethnic groups. Age Ageing. 2004 Sep;33(5):447-52. doi: 10.1093/ageing/afh135. Epub 2004 Jun 24. PMID 15217776
- [Background] Borson S, Scanlan JM, Watanabe J, Tu SP, Lessig M. Simplifying detection of cognitive impairment: comparison of the Mini-Cog and Mini-Mental State Examination in a multiethnic sample. J Am Geriatr Soc. 2005 May;53(5):871-4. doi: 10.1111/j.1532-5415.2005.53269.x. PMID 15877567
- [Background] Wilson PW, D'Agostino RB, Levy D, Belanger AM, Silbershatz H, Kannel WB. Prediction of coronary heart disease using risk factor categories. Circulation. 1998 May 12;97(18):1837-47. doi: 10.1161/01.cir.97.18.1837. PMID 9603539
- [Background] Burke LE, Styn MA, Glanz K, Ewing LJ, Elci OU, Conroy MB, Sereika SM, Acharya SD, Music E, Keating AL, Sevick MA. SMART trial: A randomized clinical trial of self-monitoring in behavioral weight management-design and baseline findings. Contemp Clin Trials. 2009 Nov;30(6):540-51. doi: 10.1016/j.cct.2009.07.003. Epub 2009 Aug 7. PMID 19665588
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Riegel B, Moser DK, Powell M, Rector TS, Havranek EP. Nonpharmacologic care by heart failure experts. J Card Fail. 2006 Mar;12(2):149-153. doi: 10.1016/j.cardfail.2005.10.004. PMID 16520265
- [Background] Romanelli J, Fauerbach JA, Bush DE, Ziegelstein RC. The significance of depression in older patients after myocardial infarction. J Am Geriatr Soc. 2002 May;50(5):817-22. doi: 10.1046/j.1532-5415.2002.50205.x. PMID 12028166
- [Background] Ziegelstein RC, Fauerbach JA, Stevens SS, Romanelli J, Richter DP, Bush DE. Patients with depression are less likely to follow recommendations to reduce cardiac risk during recovery from a myocardial infarction. Arch Intern Med. 2000 Jun 26;160(12):1818-23. doi: 10.1001/archinte.160.12.1818. PMID 10871976
- [Background] DiMatteo MR, Giordani PJ, Lepper HS, Croghan TW. Patient adherence and medical treatment outcomes: a meta-analysis. Med Care. 2002 Sep;40(9):794-811. doi: 10.1097/00005650-200209000-00009. PMID 12218770
- [Background] Kravitz RL, Hays RD, Sherbourne CD, DiMatteo MR, Rogers WH, Ordway L, Greenfield S. Recall of recommendations and adherence to advice among patients with chronic medical conditions. Arch Intern Med. 1993 Aug 23;153(16):1869-78. PMID 8250648
- [Background] Sherbourne CD, Stewart AL. The MOS social support survey. Soc Sci Med. 1991;32(6):705-14. doi: 10.1016/0277-9536(91)90150-b. PMID 2035047
- [Background] Frediani JK, Reilly CM, Higgins M, Clark PC, Gary RA, Dunbar SB. Quality and adequacy of dietary intake in a southern urban heart failure population. J Cardiovasc Nurs. 2013 Mar-Apr;28(2):119-28. doi: 10.1097/JCN.0b013e318242279e. PMID 22343212
- [Background] Schakel SF. Maintaining a nutrient database in a changing marketplace: Keeping pace with changing food products-- A research perspective. Journal of Food Composition and Analysis 2001;14:315-322.
- [Background] Heil DP. Predicting activity energy expenditure using the Actical activity monitor. Res Q Exerc Sport. 2006 Mar;77(1):64-80. doi: 10.1080/02701367.2006.10599333. PMID 16646354
- [Background] Revicki DA, Israel RG. Relationship between body mass indices and measures of body adiposity. Am J Public Health. 1986 Aug;76(8):992-4. doi: 10.2105/ajph.76.8.992. PMID 3728773
- [Background] Tothill P, James Hannan W. Dual-energy X-ray absorptiometry measurements of fat and lean masses in subjects with eating disorders. Int J Obes Relat Metab Disord. 2004 Jul;28(7):912-9. doi: 10.1038/sj.ijo.0802536. PMID 15098016
- [Background] Pickering TG, Hall JE, Appel LJ, Falkner BE, Graves JW, Hill MN, Jones DH, Kurtz T, Sheps SG, Roccella EJ; Council on High Blood Pressure Research Professional and Public Education Subcommittee, American Heart Association. Recommendations for blood pressure measurement in humans: an AHA scientific statement from the Council on High Blood Pressure Research Professional and Public Education Subcommittee. J Clin Hypertens (Greenwich). 2005 Feb;7(2):102-9. doi: 10.1111/j.1524-6175.2005.04377.x. No abstract available. PMID 15722655
- [Background] Panz VR, Raal FJ, Paiker J, Immelman R, Miles H. Performance of the CardioChek PA and Cholestech LDX point-of-care analysers compared to clinical diagnostic laboratory methods for the measurement of lipids. Cardiovasc J S Afr. 2005 Mar-Apr;16(2):112-7. PMID 15915279
- [Background] Shemesh T, Rowley KG, Shephard M, Piers LS, O'Dea K. Agreement between laboratory results and on-site pathology testing using Bayer DCA2000+ and Cholestech LDX point-of-care methods in remote Australian Aboriginal communities. Clin Chim Acta. 2006 May;367(1-2):69-76. doi: 10.1016/j.cca.2005.11.014. Epub 2006 Jan 4. PMID 16388790
- [Background] Jain A, Persaud JW, Rao N, Harvey D, Robertson L, Nirmal L, Nirmal D, Thomas M, Mikhailidis DP, Nair DR. Point of care testing is appropriate for National Health Service health check. Ann Clin Biochem. 2011 Mar;48(Pt 2):159-65. doi: 10.1258/acb.2010.010195. Epub 2011 Feb 25. PMID 21355015
- [Background] Nam S, Han HR, Song HJ, Song Y, Kim KB, Kim MT. Utility of a point-of-care device in recruiting ethnic minorities for diabetes research with community partners. J Health Care Poor Underserved. 2011 Nov;22(4):1253-63. doi: 10.1353/hpu.2011.0117. PMID 22080707
- [Background] Westlake C, Evangelista LS, Stromberg A, Ter-Galstanyan A, Vazirani S, Dracup K. Evaluation of a Web-based education and counseling pilot program for older heart failure patients. Prog Cardiovasc Nurs. 2007 Winter;22(1):20-6. doi: 10.1111/j.0889-7204.2007.05703.x. PMID 17342002
- [Background] Stepleman L, Rutter MC, Hibbard J, Johns L, Wright D, Hughes M. Validation of the patient activation measure in a multiple sclerosis clinic sample and implications for care. Disabil Rehabil. 2010;32(19):1558-67. doi: 10.3109/09638280903567885. PMID 20590506
- [Background] Kyung Rim Shin, Mi Young Kim, Seung Eun Chung. Methods and strategies utilized in published qualitative research. Qual Health Res. 2009 Jun;19(6):850-8. doi: 10.1177/1049732309335857. PMID 19429769
- [Background] Goldstein DJ. Beneficial health effects of modest weight loss. Int J Obes Relat Metab Disord. 1992 Jun;16(6):397-415. PMID 1322866
- [Derived] Cacciata M, Candelaria D, Reyes AT, Serafica R, Hildebrand JA, Santa Maria A, Lee JA, Stromberg A, Evangelista LS. Digital Health Technologies to Promote Healthy Eating and Physical Activity and Reduce Risk Factors for Cardiovascular Disease in Older Adults: A Pilot Study. J Cardiovasc Nurs. 2025 Sep-Oct 01;40(5):475-485. doi: 10.1097/JCN.0000000000001184. Epub 2025 Mar 10. PMID 40059110
- [Derived] Candelaria D, Cacciata M, Serafica R, Reyes AT, Lee JA, Hildebrand JA, Sta Maria A, Stromberg A, Evangelista LS. Patient activation improves with a multi-component personalized mHealth intervention in older patients at risk of cardiovascular disease: a pilot randomized controlled trial. Eur J Cardiovasc Nurs. 2025 Mar 3;24(2):316-322. doi: 10.1093/eurjcn/zvae159. PMID 39756174
- See also: My Fitness Pal — https://www.myfitnesspal.com/